CLINICAL TRIAL: NCT05576090
Title: Mindful Awareness Practices vs. Sleep Education: Improving Sleep Quality During the Transition to College
Brief Title: UCLA REST Study (REsearch on Sleep Techniques)
Acronym: REST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Julienne Bower, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-000229
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disturbance; Inflammation; Psychosocial Functioning
Keywords: Sleep; Adolescents; Mindfulness Meditation; Inflammation
MeSH Terms: conditions — Parasomnias; Inflammation | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation (Experimental): Half of the subjects will be randomly assigned to participate in the Mindfulness Meditation intervention. This class will meet once a week, for two hours, over the course of six weeks.
  Interventions: Behavioral: Mindfulness Meditation
- Sleep Education (Active Comparator): Half of the subjects will be randomly assigned to participate in the Sleep Education intervention. This class will meet once a week, for two hours, over the course of six weeks.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Mindfulness Meditation — The mindful awareness practices (MAPS) for Sleep intervention is based on an institutional program developed by the Mindful Awareness Research Center (MARC) at UCLA. This intervention includes educational and behavioral content related to sleep, including the importance of regularity of sleep schedules, minimizing noise and light, and reducing caffeine use later in the day. Each session provides structured training and exercises in mindfulness, including formal meditation practices and strategies for the daily informal use of mindfulness, as well as opportunity for questions and group discussion. Home practice is a key component of MAPs and is particularly important for addressing sleep disturbance. Participants will be instructed to practice mindfulness techniques on a daily basis, beginning with five minutes and increasing to 20 minutes, with practice prior to bedtime, and to practice at night if they awake and cannot return to sleep.
  Other Names: MAPS for Sleep Intervention
  Arms: Mindfulness Meditation
Behavioral: Sleep Education — The Sleep Education intervention provides education and behavioral content based on the National Institutes of Health and National Sleep Foundation tips for better sleep (e.g., changing poor sleep habits and establishing a bedtime routine). Each session provides didactic instruction, review of behavioral techniques, and opportunity for questions. Homework includes practicing sleep hygiene and weekly reading. Key components of the intervention include information about sleep biology, characteristics of healthy and unhealthy sleep, sleep problems, stress biology and stress reduction, self-monitoring of sleep behavior, relaxation methods for improving sleep, and weekly behavioral sleep hygiene strategies.
  Arms: Sleep Education

SUMMARY:
Sleep disturbance has a range of negative effects on psychosocial and biological processes important for academic and social success as well as mental and physical health among adolescents and young adults. Limited, inconsistent, and poor quality sleep lead to anxiety, depressive feelings, loneliness, and fatigue over time. These symptoms, in turn, interfere with the ability to get a good night's rest. Sleep disruption can also upregulate inflammatory processes during the years of adolescence and young adulthood in ways that can create risk for the development of chronic health conditions (e.g., diabetes, depression, cardiovascular disease) in later adulthood. Sleep, however, is also a modifiable health behavior, leading many institutions to embark upon efforts to improve the sleep of their students. The challenge is to identify programs and interventions that can simultaneously improve sleep, be delivered at scale, and be easily completed by students. UCLA has developed and validated a group-based mindfulness intervention, Mindful Awareness Practices (MAPs), that has demonstrated beneficial effects on sleep in adults and may offer a promising, scalable approach for reducing sleep disturbance and improving associated psychological and biological outcomes in college students. However, this approach requires validation in this population relative to sleep education programs, which increasingly dominate the college landscape. To address this important public health problem, the investigators propose to conduct a single site, two-arm, parallel group randomized controlled trial to test the efficacy of the validated, group-based, six-week MAPs intervention vs. sleep education, an active time and attention matched control condition, for first and second year undergraduate students who report poor sleep at this critical transition year. The investigators are aiming to enroll approximately 240 participants. Participants will complete questionnaires, provide blood samples for immune analysis and will be provided with wrist actigraphs to wear for 7 days, in order to collect objective measurements of sleep at pre- and post-intervention visits, and at a 3-month follow-up visit. Additional follow-up assessments will take place at 6-month, and 12-month post-intervention to evaluate persistence of effects.

DETAILED DESCRIPTION:
Sleep disruption during college presents a significant public health concern, with studies documenting clinically-significant sleep disruption in 40-60% of college students. Poor sleep contributes to rising anxiety, depression, and loneliness as well as declining positive affect, motivation, and sense of purpose faced by many students as they attempt to navigate a successful path through college. Disrupted sleep also negatively impacts physical health, in part through up-regulating inflammatory processes that have acute and more chronic effects on a variety of health-related outcomes.

Overview: This single-site, two-arm, parallel group randomized controlled trial will evaluate the efficacy of a mindfulness-based intervention for sleep disturbance (Mindful Awareness Practices for Sleep (MAPs)) relative to an active sleep education control condition for first and second-year undergraduate students with sleep disturbance. Both interventions will be delivered in a group format once per week for six weeks, in the students' residential halls, and led by experienced instructors following manualized protocols. Groups will be conducted in the evenings at standardized times (weeks 3-8) during the 10-week quarter to avoid conflict with final exams. Assessments will be conducted pre- and post-intervention and at 3, 6, and 12-month post-intervention follow-ups to evaluate persistence of effects. All assessments will be conducted during the academic year.

Participants: Study participants will be first year and second year undergraduate students at UCLA who endorse sleep disturbance as determined by a score of 8 or higher on the Insomnia Severity Index (ISI). They will be recruited in cohorts of 40-50 and randomized 1:1 to one of the two study arms (20-25 students per group, the optimal group size for the MAPs intervention). Participants will complete questionnaires and blood collection at in-person assessments conducted before and after the six-week intervention and at a 3-month post-intervention follow-up. Longer-term effects on self-reported outcomes will be assessed at 6- and 12-months post-intervention. Of note, the three follow-up assessments were scheduled to avoid the summer months given the focus on improving sleep in the college context.

Eligibility Screening: Potential participants will be directed to contact the study coordinator via email, phone, or a secure online signup form. The coordinator will then contact potential participants by phone to confirm eligibility criteria. The ISI will be administered to screen for current insomnia. Those who score an "8" or above, indicating at least sub-threshold levels of sleep disturbance, will be considered eligible for study participation. The 4-item Patient Health Questionnaire (PHQ4) survey will be used to screen for a diagnosis of a current mood or anxiety disorder. The 4-item PHQ-4 screening measure provides a good measure of "caseness" for both anxiety and depression that has been validated in college samples. If a potential subject scores a "3" on either subscale, the study coordinator will administer the 8-item Patient Health Questionnaire (PHQ8) for depression or the 7-item Generalized Anxiety Disorder (GAD-7) for anxiety, to determine the severity. If the potential participant scores "15" or more on either scale, they will be referred to the UCLA Counseling and Psychological Services (CAPS). Screening will continue until there are 45-50 participants who are eligible, interested, and available to participate in the next cohort.

Enrollment and Baseline Assessment (T1). All students who are determined to be eligible will be scheduled for an in-person, baseline assessment (T1) at the UCLA Health Psychology Laboratory (HPL). The Institutional Review Board (IRB) approved consent form will be reviewed and signed. A pre-intervention online survey will also be completed during this initial in-person visit. The survey will consist of the following scales: Background demographic and medical characteristics, health behaviors, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI), Anxiety and Preoccupation with Sleep (APSQ), Center for Epidemiological Studies-Depression (CES-D), Generalized Anxiety Disorder-7 (GAD-7), Multi-dimensional Fatigue Symptom Inventory Short Form (MFSI-SF), Perceived Stress Scale (PSS), UCLA Loneliness Scale, Positive and Negative Affect Scale (PANAS-X, positive affect subscales), Mental Health Continuum-Short Form (MHC-SF), Mindfulness scale (FFMQ), Self-Compassion Scale (self-kindness subscale), and the Rumination and Reflection Questionnaire (rumination subscale).

Participants will provide blood samples for immune evaluation using the Tasso OnDemand device, which allows self-collection of a single capillary blood sample and does not require venipuncture. The Tasso device sticks to the skin with a light adhesive. When the button is pressed, a vacuum forms and a lancet pricks the surface of the skin. The vacuum draws blood out of the capillaries and into a sample pod attached to the bottom of the device. Participants will watch a demonstration video during their baseline assessment visit, and then use the device to collect a blood sample. Approximately 1/8th of a teaspoon of blood will be drawn at each in-person assessment.

Participants will be provided with a wrist actigraph (Micro Motionlogger Sleep Watch, Ambulatory Monitoring, Inc.; Ardsley, NY) to wear on their non-dominant hand for seven consecutive 24-hour periods. They will be instructed to keep it on at all times, removing only for bathing. Participants will be instructed to press the event marker on the actigraph to indicate when they: 1) turn off the lights to go to sleep at night, 2) get out of bed in the middle of the night, such as to use the bathroom, 3) get out of bed in the morning, and 4) begin and end daytime naps. The software package Action 4 (Ambulatory Monitoring, Inc.; Ardsley, NY) will be used to code and score the actigraphy data, and established algorithms will be used to provide estimates of parameters such as sleep duration, sleep onset latency, efficiency, daily variability, and wakenings after sleep onset.

Assessments will be scheduled in the morning to control for diurnal variations in immune parameters. Baseline visits will be conducted in the 2-week period before intervention onset.

Randomization: Following baseline assessment, participants will be randomized to one of the two study conditions. Participants will be stratified based on gender (female/male/non-binary or other) and ISI score (less than 14/14 and above) and then randomized with 1:1 allocation to the two conditions. The randomization sequence will be generated using the PLAN procedure in SAS 9.4 and uploaded into REDCap. The study coordinator will use the REDCAP "Randomize" procedure to determine the participant's assigned condition. The coordinator will inform the participants of their assigned condition and provide information on the intervention.

Interventions: Both interventions will be held in private rooms in the residential part of the UCLA campus, close to student living quarters. Group sessions will be conducted in the evenings and scheduled to occur mid-way through the quarter (weeks 3-8 of the 10-week quarter) to minimize conflict with classes and exam periods.

Mindful Awareness Practices for Sleep (MAPs): Participants assigned to this condition will be asked to attend two-hour group sessions once a week for six weeks. The MAPs intervention is based on an institutional program developed by the Mindful Awareness Research Center (MARC) at UCLA and adapted to specifically address sleep disturbance. The MAPs program is similar to other mindfulness-based interventions in its general focus on cultivating mindfulness, but takes a more practical and accessible approach that focuses specifically on the practice of mindfulness and its application in everyday life (as compared to the focus on stress and stress reduction in mindfulness-based stress reduction). Key components of the intervention include development of bodily awareness, managing pain, working with difficult thoughts and feelings, cultivating positive emotions and loving kindness, and relational mindfulness practices. The MAPs curriculum will be implemented by trained instructors who will receive specialized training in delivery of the study-specific protocol and will be overseen by Diana Winston, Director of Education at the Mindful Awareness Research Center.

Sleep Education (SE): Participants assigned to this condition will be asked to attend a two-hour group session once a week for 6 weeks. This program is based on the sleep education program used by Dr. Michael Irwin and colleagues, and matches the MAPs condition for time, attention, group interaction, and expectancy of benefit. The SE intervention provides education and behavioral content based on the National Institutes of Health and National Sleep Foundation tips for better sleep (e.g., changing poor sleep habits and establishing a bedtime routine).The standardized program will be implemented by trained health educators who will receive specialized training in delivery of the study-specific protocol with oversight by Co-I Dr. Michael Irwin.

Immediate Post-Intervention Assessment (T2): This in-person visit will be scheduled to occur within 2 weeks after the conclusion of the study interventions at the UCLA HPL and will include completion of study questionnaires, collection of blood samples, and 7 days of actigraphy.

3-, 6-, and 12-month Follow-up Assessments (T3,T4,T5). All participants will be asked to complete follow-up assessments at 3 months (T3), 6 months (T4), and 12 months (T5) post-intervention. The T3 assessment will be conducted at the UCLA HPL and will include completion of questionnaires, blood collection, and 7 days of actigraphy. T4 and T5 assessments will involve completion of online study questionnaires only (no blood draw or actigraphy). This assessment schedule will allow the investigators to capture short- and long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* First or second year undergraduate student at UCLA
* Ages 18-22 years old
* Must live in the residential halls on UCLA campus
* Must have a score of 8 or above on the Insomnia Severity Index (ISI), indicating at least sub-threshold levels of sleep disturbance.

Exclusion Criteria

* Current diagnosis of mood or anxiety disorder as determined by the PHQ-8 or by the GAD-7 if score "15" or more on either measure
* Presence of medical conditions or use of medications that may influence sleep or inflammation (e.g., autoimmune disorder)
* Previous or current formal instruction in mindfulness meditation (e.g., MAPs, MBSR) or current sleep education program

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in sleep quality from baseline to post-intervention on the Pittsburgh Sleep Quality Index (PSQI) | Baseline and post-intervention; 3, 6, and 12-month follow-up
  The PSQI includes 19 items, yielding seven dimensions of sleep: duration, disturbance, latency, daytime dysfunction, efficiency, quality, and sleeping medication use. Following standard procedure, we will obtain the PSQI global score by summing across all seven components. Each component has a maximum score of three points; the highest possible global score is 21. Higher PSQI global scores indicate poorer quality, with scores above 5 suggesting clinically-significant sleep disturbance. Our main analyses of the primary outcome will focus on the PSQI global score at post-intervention. Follow-up, exploratory analyses will examine whether observed effects are unique to any of the seven separate subscales of the PSQI, and whether there are intervention effects at the 3, 6, and 12-month post-intervention follow-ups.

SECONDARY OUTCOMES:
Change in insomnia severity from baseline to post-intervention on the Insomnia Severity Index (ISI) | Baseline and post-intervention; 3, 6, and 12-month follow-up
  The ISI consists of 7 items which are summed for a total score (range: 0-28) with higher scores indicating greater insomnia severity. Scores of 8-14 indicate subthreshold insomnia, while scores of 15-28 indicate clinical insomnia.
Change in actigraphy-based objective sleep measures from baseline to post-intervention. | Baseline and post-intervention; 3-month follow-up
  We will obtain objective estimates of sleep using wrist actigraphy. At the baseline assessment prior to randomization (T1) and at T2 and T3, participants will be provided with a wrist actigraph (Micro Motionlogger Sleep Watch, Ambulatory Monitoring, Inc.; Ardsley, NY) to wear on their non-dominant hand for seven consecutive 24-hour periods. The software package Action 4 (Ambulatory Monitoring, Inc.; Ardsley, NY) will be used to code and score the actigraphy data, and established algorithms will be used to provide estimates of parameters such as sleep duration, sleep onset latency, efficiency, daily variability, and wakenings after sleep onset.
Change in depressive symptoms from baseline to post-intervention on the Center for Epidemiological Studies Depression Scale (CES-D) | Baseline and post-intervention; 3, 6, and 12-month follow-up
  The 20-item CES-D is a measure of depression symptom severity, with higher scores (range: 0-60) indicating greater depressive symptoms
Change in anxiety from baseline to post-intervention on the Generalized Anxiety Disorder- 7 (GAD-7). | Baseline and post-intervention; 3, 6, and 12-month follow-up
  Symptoms of anxiety will be measured via the 7-item GAD-7. Higher scores (range: 0-21) indicate greater severity of symptoms
Change in perceived stress from baseline to post-intervention on the Perceived Stress Scale (PSS). | Baseline and post-intervention; 3, 6, and 12-month follow-up
  Perceived stress will be measured via the 10-item PSS (range: 0-40). Higher scores indicate greater perceived stress levels.
Change in loneliness from baseline to post-intervention on the UCLA Loneliness Scale | Baseline and post-intervention; 3, 6, and 12-month follow-up
  Loneliness will be measured via the 3-item UCLA Loneliness Scale (range: 3-9). Higher scores indicate greater loneliness
Change in fatigue from baseline to post-intervention on the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) general fatigue subscale. | Baseline and post-intervention; 3, 6, and 12-month follow-up
  Fatigue will be measured via the MFSI-SF general fatigue subscale. This subscale consists of 6 items which are scored for a total sum (range: 0-24). Higher scores indicate greater general fatigue.
Change in positive affect from baseline to post-intervention on the Positive and Negative Affect Schedule (PANAS-X) | Baseline and post-intervention; 3, 6, and 12-month follow-up
  Positive affect will be assessed using the following subscales on the PANAS-X: the 10-item positive affect subscale, the 3-item serenity subscale and the 8-item joviality subscale. Higher scores indicate higher feelings of positive affect (range: 21-105).
Changes in psychological well-being from baseline to post-intervention on the Mental Health Continuum-Short Form (MHC-SF) | Baseline and post-intervention; 3, 6, and 12-month follow-up
  The 14-item MHC-SF is comprised of three empirically derived subscales: the 3-item Emotional Well-Being Subscale, the 6-item Psychological Well-Being Subscale, and the 5-item Social Well-Being Subscale. Higher scores on each subscale, and the total score overall (range: 0-56), indicate greater well-being.
Changes in inflammation from baseline to post-intervention | Baseline, at 8 weeks and at 20 weeks
  Pro- inflammatory gene expression will be measured through a set of 19 pre-specified pro-inflammatory gene transcripts that have previously been shown to be upregulated in the context of chronic stress and downregulated by the mindfulness meditation intervention. In addition, protein markers of inflammation will be assessed, including IL-6, IL-8, IL-10, TNF-α, IFN-γ, and CRP.
Change in worry about sleep from baseline to post-intervention on the Anxiety and Preoccupation with Sleep Questionnaire (APSQ) | Baseline and post-intervention; 3, 6, and 12-month follow-up
  The APSQ has 10 items that can be summed for a total score (range: 10-100). There are also 2 subscales: 6-items determine worries about the consequences of poor sleep and 4-items assess worries about the uncontrollability with sleep, each of which can be summed for a subscale total score. Higher scores indicate greater anxiety and preoccupation about sleep difficulties.
Change in mindfulness from baseline to post-intervention on the 15-item Five Facet Mindfulness Questionnaire (FFMQ-15) | Baseline and post-intervention; 3, 6, and 12-month follow-up
  The FFMQ-15 is comprised of 5 facets: observing, describing, acting with awareness, non-judgment and non-reactivity, along with an overall mindfulness score. The total FFMQ can be divided by 15 to get an average item score. Scores represent a spectrum of mindfulness.
Change in self-kindness from baseline to post-intervention on the Self-Compassion Scale. | Baseline and post-intervention; 3, 6, and 12-month follow-up
  Self-kindness will be measured via the 5-item self-kindness subscale from the Self-Compassion Scale. A self-kindness score is computed by calculating the mean of the 5-items. Higher scores indicate greater self-kindness.
Change in rumination from baseline to post-intervention on the Rumination and Reflection Questionnaire (RRQ) | Baseline and post-intervention; 3, 6, and 12-month follow-up
  Rumination will be measured via the 6-item rumination subscale from the Rumination and Reflection Questionnaire. Higher scores indicate more rumination.

CONTACTS AND LOCATIONS:
Overall Officials: Julienne E Bower, Ph.D., Principal Investigator — University of California, Los Angeles; Andrew Fuligni, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any individual participant data (IPD) with any other researchers. Data will be reported in group form to prevent personal identification of participants. When the research has been completed, the data will be stored in a secured area of a private, locked research office. Any personal identifiers and/or codes linking the data to personal identifiers will be kept on a separate computer with password protection for reference and for future research. All personal identifiers will be kept confidential. Only identified members of the research team and the P.I. will have access to the data, identifiers and/or codes. Data with subject identifiers will not be released to any agency or persons.